CLINICAL TRIAL: NCT04869202
Title: Fetomaternal Outcomes of Pregnancies Complicated by COVID-19 Infection; Prospective Study in a Tertiary University Hospital
Brief Title: Covid-19 Infection in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, University of Jordan
Other Study IDs: Jordan University Hospital
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Perinatology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 test — Naso-pharyngeal swab test

SUMMARY:
Prospective study of both maternal and fetal outcomes of those pregnancies that were complicated by COVID-19 infection at various gestational ages. The follow up will be from the time the diagnosis was made till discharge of the mother and her baby from the hospital.

DETAILED DESCRIPTION:
Pregnancies that have a confirmed covid-19 infection by nasopharyngeal swab whether taken at our laboratory or confirmed at private or Ministry of health (MOH) laboratories will be followed up till delivery and discharge from the hospital.

They will be followed up for hospitalization, intensive care unit (ICU) admission, any complications (organ failure, DIC, renal failure, septic shock), intubation, mortality, miscarriage, congenital malformations, intra-uterine growth restriction (IUGR), oligohydramnios, spontaneous preterm birth, mode of delivery, birth weight, APGAR score at 1 and 5 minutes, neonatal infection with covid-19, neonatal ICU admission and breast feeding. Those patients will be followed up prospectively at our hospital and those with missed follow up and delivered outside our unit will be contacted to bring all the above-mentioned parameters. There will be no exclusion of cases.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women infected with COVID-19
Study Population: Pregnant women who contract COVID-19 virus infection during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
feto-maternal outcome | 1 year
  fetal and maternal consequences of the infection

CONTACTS AND LOCATIONS:
Overall Officials: Asma Basha, Study Director — The University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided